CLINICAL TRIAL: NCT04602351
Title: Communication in ICU During COVID-19: Multinational, Multicentric Cross-sectional Survey (ComICU)
Brief Title: Communication in ICU During COVID-19
Status: Completed | Type: Observational
Sponsor: NMC Specialty Hospital (Other)
Responsible Party: Principal Investigator, Prashant Nasa, Head Critical Care Medicine, NMC Specialty Hospital
Other Study IDs: ComICU
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: COVID-19; Severe Acute Respiratory Syndrome Coronavirus 2; Severe Acute Respiratory Syndrome
Keywords: Communication in ICU; Doctor-family members communication; Informed consent
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Communication — policies on communication and informed consent in ICU

SUMMARY:
This study explores the actual situation of communication during the Coronavirus disease 2019 (COVID-19) pandemic in the South Asia and Middle East region. The purpose is to assess the effect of the limited visitor policy during the COVID-19 pandemic, on the pattern of interaction of critically ill patients to their kin/ guardian and doctor-family members communication.

Primary objective of this study are as follows:

1. Explore the changes in communication pattern with limited contact during the COVID-19 pandemic.
2. Assess the methods of informed consent in Intensive care units (ICUs) during the same period

DETAILED DESCRIPTION:
An observational, cross-sectional, web-based questionnaire survey, with multi-centre involvement across hospitals in the South Asia and middle-east region. The questionnaire consists of two sections. Section one obtains information from participants regarding communication and visiting practices in ICU during pre-COVID-19 era, and the Section two obtains information regarding the policy changes if any during the COVID-19 pandemic in regards to safety of healthcare workers (HCWs) and public.

In order to obtain the largest representation of South Asia and Middle East ICUs, a network of research doctors as facilitators from each country is created. The role of the facilitators is to contact and recruit adult ICUs within their country. Each facilitator contacts the hospitals (public and private), creating a network of collaborating doctors/nurses (participants) from those hospitals who expressed their willingness to participate.

Data collection: a web based Google Forms with online access will be used Only one entry per ICU will be collected during the study. Statistic analysis: a descriptive analysis is planned for the general characteristics of the participating units and the study population.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ICUs,
2. New created COVID-19 ICUs during the pandemic

Exclusion Criteria:

1. Paediatric ICU
2. Neonatal ICU

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU communication teams across South Asian and Middle East Region
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Changes in the pattern of family members visiting process | 12 months
  Using a questionnaire the changes in visiting policy for family members or friends will be recorded from last year (before COVID-19 pandemic).
  This will include, visiting policy, visiting hours and their change after pandemic at the time of study (November 2020).
Changes in process of communication between health care workers(HCWs) and family members | 12 months
  Through a questionnaire, the process of communication between HCWs and family members or friends before pandemic (November 2019) and November 2020 will be recorded.
  This will include the responsible HCW for communication, place of communication and method of communication (in person versus electronic)

SECONDARY OUTCOMES:
Changes in process of informed consent in ICU | 12 months
  Through a questionnaire, the process of informed consent for procedures and end of life (EOL) or do not attempt to resuscitation (DNAR) in ICU will be collected and its change in last 12 months (from November 2019 to November 2020)

CONTACTS AND LOCATIONS:
Locations (1):
- NMC Specialty Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared to ensure confidentiality and privacy of participating Institution.

REFERENCES:
- [Background] Back A, Tulsky JA, Arnold RM. Communication Skills in the Age of COVID-19. Ann Intern Med. 2020 Jun 2;172(11):759-760. doi: 10.7326/M20-1376. Epub 2020 Apr 2. PMID 32240282
- [Background] Azoulay E, Kentish-Barnes N. A 5-point strategy for improved connection with relatives of critically ill patients with COVID-19. Lancet Respir Med. 2020 Jun;8(6):e52. doi: 10.1016/S2213-2600(20)30223-X. Epub 2020 May 4. No abstract available. PMID 32380024
- [Background] Rubinelli S, Myers K, Rosenbaum M, Davis D. Implications of the current COVID-19 pandemic for communication in healthcare. Patient Educ Couns. 2020 Jun;103(6):1067-1069. doi: 10.1016/j.pec.2020.04.021. No abstract available. PMID 32451002
- [Result] van Beusekom I, Bakhshi-Raiez F, de Keizer NF, Dongelmans DA, van der Schaaf M. Reported burden on informal caregivers of ICU survivors: a literature review. Crit Care. 2016 Jan 21;20:16. doi: 10.1186/s13054-016-1185-9. PMID 26792081
- [Result] Cicekci F, Duran N, Ayhan B, Arican S, Ilban O, Kara I, Turkoglu M, Yildirim F, Hasirci I, Karaibrahimoglu A, Kara I. The communication between patient relatives and physicians in intensive care units. BMC Anesthesiol. 2017 Jul 17;17(1):97. doi: 10.1186/s12871-017-0388-1. PMID 28716040